CLINICAL TRIAL: NCT01267994
Title: A Phase I/II Open-label Study of the Effects of Anakinra in Corticosteroid-resistant Subjects With Autoimmune Inner Ear Disease
Brief Title: A Clinical Trial of Anakinra for Steroid-Resistant Autoimmune Inner Ear Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andrea Vambutas (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Andrea Vambutas, Professor of Otolaryngology & Molecular Medicine, Northwell Health
Organization: Northwell Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21DC011827-01 (NIH); R33DC011827 (NIH)
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Sensorineural Hearing Loss; Autoimmune Inner Ear Disease
Keywords: Steroid; Steroid-Resistant; Autoimmune Inner Ear Disease; Immune Mediated Hearing Loss; Sudden Sensorineural Hearing Loss; Meniere's Disease; Autoimmune; Hearing
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Sudden; Meniere Disease | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm-Open Label (Experimental): Single Arm-Open Label use of Anakinra
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — 100mg of anakinra administered by a subcutaneous injection for 84 consecutive days.
  Other Names: Kineret

SUMMARY:
The purpose of this study is to determine if Anakinra (an interleukin-1 receptor antagonist) can improve hearing thresholds in those patients with Autoimmune Inner Ear Disease (AIED) that did not respond to oral steroid therapy for a sudden decline in hearing. The patients to be enrolled will have recently completed a course of oral steroids and demonstrated no change in their audiometric thresholds following corticosteroid therapy.

DETAILED DESCRIPTION:
Patients with immune mediated hearing loss (also known as autoimmune hearing loss) are typically treated with corticosteroids. Of those treated, approximately 60% respond, however, that response may be lost over time. Other therapies use to date have proven largely ineffectual in improving hearing. This study proposes a phase I open label clinical trial of Anakinra for corticosteroid-resistant patients to determine if this therapy is efficacious in hearing restoration.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral sensorineural hearing loss with an active decline in hearing in one ear
* No audiometric improvement with 28-30 days of oral prednisone or other corticosteroid, including an initial dose of 60mg per day for 14 days
* Enrollment within 14 days of completion of corticosteroid therapy
* Age 13 years and older
* No evidence of neutropenia (low white blood cell count)
* No evidence of retrocochlear pathology (ie. acoustic neuroma/vestibular schwannoma)
* May have concurrent, systemic autoimmune disease

Exclusion Criteria:

* Age over 75, or less than 13
* Neutropenia
* Renal insufficiency
* Pregnant females
* Unilateral hearing loss
* Patients with any immunodeficiency syndrome
* Patients receiving methotrexate or any TNF (tumor necrosis factor) antagonist therapy
* Patients with chronic infections
* Patients treated for a malignancy within the past 3 years
* Patients with a latex allergy
* Patients with an inner ear anomaly
* Patients with retrocochlear pathology

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vambutas, MD, Principal Investigator — Northwell Health
Locations (1):
- North Shore-LIJ Hearing and Speech Center, New Hyde Park, New York, United States

REFERENCES:
- [Result] Vambutas A, Lesser M, Mullooly V, Pathak S, Zahtz G, Rosen L, Goldofsky E. Early efficacy trial of anakinra in corticosteroid-resistant autoimmune inner ear disease. J Clin Invest. 2014 Sep;124(9):4115-22. doi: 10.1172/JCI76503. Epub 2014 Aug 18. PMID 25133431
- See also: Clinical trials at the Feinstein Institute for Medical Research — http://www.feinsteininstitute.org/Feinstein/Clinical+Trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Trial: Open label, single arm trial of anakinra for corticosteroid-resistant Autoimmune Inner Ear Disease
Period: Overall Study
Arm/Group | Open Label Trial
Started | 12 (Declined to participate. n=1 Did not receive intervention due to infeciton, n=1)
Completed | 10 (Excluded from analysis, could not reach first milestone (day 28) for efficacy assessment, n=2)
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Corticosteroid-resistant AIED patients.
Groups:
- Single Arm: Patients with Autoimmune Inner Ear Disease that had <5dB hearing improvement in response to corticosteorids following 28 days of treatment
Arm/Group | Single Arm
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — 14 Non-responders, 1 elected not to participate
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 13
    More than one race | 0
    Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Potential Efficacy of Anakinra in Improving Hearing Thresholds in Corticosteroid-resistant Patients With Autoimmune Inner Ear Disease
Description: The primary endpoint is to determine whether those treated with anakinra for 84 days demonstrate an improved hearing threshold compared with their pre-anakinra-treatment threshold. Audiometric thresholds will be compared to those treated with a prolonged corticosteroid taper and those that elect for no further treatment. The durability of the response will be measured over a total of 180 days.
Time Frame: 180 days
Measure: Number; unit: responders
Arm/Group | Single Arm
Number analyzed (Participants) | 10
responders | 7

2. Secondary Outcome: Number of Serious Adverse Events Reported
Description: To assess the number of Serious Adverse Events reported in any subject that received at least one injection dose of anakinra
Time Frame: 84 days
Population: Any subject enrolled in this study who received at least 1 injection dose of anakinra
Measure: Number; unit: reported SAEs
Groups:
- Single Arm: Subject who received at least one injection of anakinra
Arm/Group | Single Arm
Number analyzed (Participants) | 12
reported SAEs | 0

ADVERSE EVENTS:
Groups:
- Single Arm: Anakinra administered for 84 consecutive days
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=12)
Injection site reactions (Skin and subcutaneous tissue disorders) | 10 — Injection site reactions
Headache (Nervous system disorders) | 4
Vertigo (Nervous system disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 2
Influenza like illness (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Psoriasis Flare (Skin and subcutaneous tissue disorders) | 1
Visual Impairment (Eye disorders) | 1 — floaters

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No